CLINICAL TRIAL: NCT04667065
Title: Evaluation of a Remotely Guided Physical Preparation by a Physical Activity Teacher Adapted With the Help of a Smartwatch Before Bronchial Cancer Surgery
Acronym: PREPACHIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PREPACHIR
Record Dates: First submitted 2020-11-25; First posted 2020-12-14 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Lung Cancer
Keywords: smartwatch, lung cancer operation, physical exercices
MeSH Terms: conditions — Lung Neoplasms | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Patient with non-small cell bronchial cancer with indication of curative surgical resection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physical activity with smartwatch before bronchial cancer surgery (Other)
  Interventions: Other: Physical activity

INTERVENTIONS:
Other: Physical activity — Physical activity with the remotely guidance of physical activity teachers

SUMMARY:
This is a study of a preoperative rehabilitation program with remotely guided high-intensity exercises by physical activity teachers adapted to a smartwatch in patients with operable lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Major patient, age ≥ 18
* Patient with non-small cell operable bronchial cancer without indication of neo-adjuvant chemotherapy
* Affiliated with a social security plan
* VEMS < 80% and/or DLCO<80%
* High-intensity training achievable for at least 10 days before surgery
* Acceptant to participate in the protocol
* Ability to follow the STIMUL program of education focused on adapted physical activity
* Have a smartphone that can download the mobile app
* have the ability to understand, read and write French

Exclusion Criteria:

* Patient unable to consent: under guardianship or curatorship
* Patient refusing surgery
* Non-operable patient due to comorbidities or unseable tumour
* Poor understanding of the smartwatch
* Severe cognitive or psychiatric disorders
* Pregnancy in progress

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Measure of VO2 max . | 1 day before surgery
  comparison of VO2 max at inclusion and one day before surgery

SECONDARY OUTCOMES:
Number of patients who used the remotely guided physical preparation | one day before surgery
maximum distance covered in the 6-minute walking t | one day before surgery
post-surgery complications | At 1 month and 3 months
number of individuals who participated in the physical activity program | one day before surgery
post surgery intubation duration | At 1 month
number of days at hospital | At 3 months
number of days with oxygen | At 1 month and 3 months
(forced expiratory volume | At 1 month and 3 months
capacity of carbon monoxide | At 1 month and 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Centre hospitalier intercommunal de Créteil, Créteil, France